CLINICAL TRIAL: NCT00842335
Title: A Multicenter, Phase 1/2, Open-Label, Dose-Escalation Study of JI-101, an Oral Angiogenesis Inhibitor, in Patients With Advanced Solid Tumors
Brief Title: A Phase 1/2, Open-Label, Dose-Escalation Study of JI-101, in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jubilant Innovation Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JI-101-001
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Advanced Solid Tumors
Keywords: solid tumors; angiogenesis inhibitor; dose escalation; maximum tolerated dose; JI-101
MeSH Terms: interventions — 1-(1-(2-amino-pyridin-4-ylmethyl)-1H-indol-4-yl)-3-(5-bromo-2-methoxyphenyl)urea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- JI-101 (Experimental)
  Interventions: Drug: JI-101

INTERVENTIONS:
Drug: JI-101 — JI-101, 50 mg capsules, will be administered daily for up to 112 days (four 28-day cycles); treatment may be extended if, in the opinion of the investigator, a patient has tolerated the treatment and appears to be benefitting from receiving study medication

SUMMARY:
The purpose of this study, the first clinical trial of JI-101, is to determine the maximum tolerated dose of JI-101 when given orally to patients with solid tumors. Safety, tolerability, pharmacokinetics, pharmacodynamics, and the effects of the drug on tumor metabolism will also be studied. JI-101 is an inhibitor of new blood vessel growth that may provide benefit to patients with solid tumors that have failed standard therapeutic regimens.

DETAILED DESCRIPTION:
JI-101 is a compound being developed for the treatment of patients with solid tumors; specifically patients for which no approved therapy or standard of care is available or have solid tumors and have failed standard of care therapy. JI-101 is an inhibitor of vascular endothelial growth factor receptor 2 (VEGFR2), platelet-derived growth factor receptor beta (PDGFRβ), and EphB4 receptor, each of which plays an important role in driving vascularization (angiogenesis and vasculogenesis) during normal development and tumorigenesis. JI-101 inhibits the growth of new blood vessels, which in turn, may slow or prevent the growth of tumors. The purpose of this open label study is to treat patients with advanced solid tumors, with increasing doses of JI-101, thereby providing information about the maximum tolerated dose (MTD). The study will also examine safety, tolerability, pharmacokinetics, pharmacodynamics, and may evaluate the effects of the drug on tumor metabolism. During this dose-escalation study, at least two patients will be dosed at each dose level (cohort). The patients must complete 21 days of dosing and safety results will be reviewed prior to any patients being assigned the next higher dose level. A continuous reassessment method will be utilized to escalate JI-101 doses between cohorts. Doses will be increased, with an anticipated high dose of 800mg per day. If the MTD is not reached, an optimal biologic dose (OBD) will be determined based on the highest doses that are tolerable with acceptable efficacy. The cohort at MTD or OBD will be expanded to include up to 30 patients with solid tumors to further explore the safety and tolerability of orally-administered JI-101.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or greater at the time of consent.
* Have solid tumors for which no approved therapy or standard of care is available or have solid tumors and have failed standard-of-care therapy.
* Have life expectancy of greater than 3 months.
* Have Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* Have organ and marrow function as defined below:

  * absolute neutrophil count ≥ 1.5 x 10^9 cells/L
  * hemoglobin ≥ 9.0 g/dL
  * platelets ≥ 75 x 10^9 cells/L
  * total bilirubin ≤ 1.5 x upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 2.5 x ULN (≤ 5 x ULN for liver metastases)
  * serum creatinine < 1.5 x ULN
  * < 500 mg urinary protein/24 hours or dipstick < 2+
* No evidence of preexisting uncontrolled hypertension as documented by two baseline blood pressure readings taken at least 1 hour apart (the baseline systolic blood pressure readings must be <140 mm Hg, and the baseline diastolic blood pressure readings must be <90 mm Hg. Patients whose hypertension is controlled by antihypertensive therapies are eligible)
* Have no clinically significant disease that poses a risk to the patient and/or would interfere with study evaluations or procedures.
* Have within normal range cardiac function as measured by twelve-lead electrocardiogram at Screening.
* Be clinically euthyroid.
* If female, must be postmenopausal (at least 1 year from last menses), or surgically sterile, or if a female patient of childbearing potential they must agree to use acceptable methods of birth control, which include local double-barrier contraceptive methods, such as cervical diaphragm plus spermicide, female condom plus spermicide, or a non-hormonal intrauterine device (IUD) plus spermicide, or systemic contraceptive methods, such as oral, injectable, transdermal or implantable hormonal contraceptives (including hormone-containing IUDs) during the study period, and for 30 days after the last dose of study drug. Female patients of childbearing potential must have a negative serum pregnancy test within the 3 days before the first study drug administration. Male patients must be surgically sterile or also agree to use acceptable methods of birth control with their female partners, and this may include use of a male condom plus spermicide. If the subject is practicing abstinence at the time of Screening, he/she must agree to use a double-barrier contraceptive method if he/she becomes sexually active.
* Be able to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Be pregnant or breastfeeding.
* Have a known history of human immunodeficiency virus (HIV) infection because the effect of JI-101 on immunosuppression and drug interactions with anti-retroviral medications is unknown.
* Have participated in an investigational drug/device/biologic study within 30 days (or within 5 half-lives of the treatment, whichever is longer) before Visit 1 or who are currently participating in another investigational drug/device/biologic study. Participation in non-interventional or observational studies is allowed.
* Have a history of cardiac abnormalities including: abnormal and clinically relevant ECGs; frequent palpitations or syncopal episodes; heart failure; hypokalemia; stroke; family history of Long QT Syndrome; acute myocardial infarction or ventricular tachyarrhythmia within the previous 12 months.
* Have used concomitant medications that prolong the QT/QTc interval within 14 days prior to Day 1.
* Have a history of significant retinopathy or any progressive eye disease that could lead to severe loss of visual acuity or visual field loss during the study period.
* Have had therapeutic reanticoagulation with heparin or heparin analogs (low molecular weight heparins) or warfarin within the past 4 weeks. Low dose warfarin (1 to 2 mg/day) is allowed for prophylaxis treatment.
* Have had major surgery, radiotherapy, chemotherapy, or cytokine therapy within 4 weeks of treatment initiation. Patients must have recovered to baseline or grade 1 from any clinically significant adverse event experienced during those prior therapies.
* Have gastrointestinal abnormalities including inability to take oral medications, malabsorption syndromes or other clinically significant GI abnormalities that may impair the absorption of JI-101 in the opinion of the Investigator.
* Have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, or psychiatric illness/social situations that would pose a risk to patient safety or that would limit compliance with study requirements.
* Have any condition that, in the opinion of the Investigator, would interfere with a patient's ability to perform the required activities of the study or would subject the patient to undue risk.
* Patients with proteinuria (patients with >2+ protein on urine dipstick) at baseline should undergo a 24-hour urine collection. Results must demonstrate <500 mg of protein in 24 hours to allow participation in the study)
* Patients with any of the following contraindications to FDG-PET can participate in the study if all of the inclusion criteria and none of the exclusion criteria are met, but these patients are excluded from FDG PET assessments:

  o Inability to remain lying down in PET scanner (for PET portion of the study).
* Absence of at least one metastatic lesion greater than or equal to 2 cm on pre-dose CT (computed tomography) scan or other radiographic imaging as defined by response evaluation criteria in solid tumors (RECIST) criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Premiere Oncology of Arizona, Scottsdale, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one clinical site in the US. First Patient Enrolled: 24 February 2009 Cut-off Date: 15 February 2011
Groups:
- JI-101: JI-101 : JI-101, 50 mg capsules, will be administered daily for up to 112 days (four 28-day cycles); treatment may be extended if, in the opinion of the investigator, a patient has tolerated the treatment and appears to be benefitting from receiving study medication
Period: Overall Study
Arm/Group | JI-101
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | JI-101
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 59.8 (9.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of JI-101
Description: The primary objective of this study was to determine the maximum tolerated dose (MTD) of JI-101 when administered orally in patients with advanced solid tumors.
  The MTD was established based on safety data from Cycle 1. Patients who completed 21 days of treatment in Cycle 1 were considered to have completed the study for the determination of MTD.
  Patients were eligible to continue treatment with JI-101 until they experienced disease progression or unacceptable treatment-related toxicity. Unacceptable treatment-related toxicity was defined as a clinically significant AE or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications, and that was attributed to JI 101.
Time Frame: 28 days (1 cycle)
Population: Full Analysis Population (FAS) or Modified Intent-to-Treat (mITT) Population: All patients enrolled into the study who received JI-101 and completed at least 21 days of dosing in Cycle 1 comprised the FAS.
  Safety Population: Included all patients who received at least one dose of study drug. This population was used for all safety analyses.
Measure: Number; unit: mg
Arm/Group | JI-101
Number analyzed (Participants) | 18
mg | 400

2. Secondary Outcome: Number of Participants Reaching Maximum Tolerated Dose
Description: Number of participants withdrawn from study due to adverse events
Time Frame: Up to 112 days (up to four 28-day cycles) or longer if the patient is benefiting from treatment
Population: Only one subject withdrew due to an adverse event.
Measure: Number; unit: participants
Groups:
- All Subjects: The starting dose of JI-101 for patients in the first cohort was 100 mg QD. All patients took JI-101 without food on Day 0, with a high fat meal on Day 2, and with a regular diet on Day 3 onwards. Patients in the first three cohorts were dosed QD. Based on PK characteristics observed from the first eight patients (Cohort 1, Cohort 2, and Cohort 3), subsequent cohorts were dosed BID.
  After the first eight patients, the combined PK profiles of the enrolled patients were studied. These assessments indicated that the PK profile for JI-101 supported BID dosing. Therefore, BID dosing was administered to patients who enrolled in the study following the effective date of Protocol
Arm/Group | All Subjects
Number analyzed (Participants) | 18
participants | 18

3. Secondary Outcome: Overall Clinical Response by Cycle
Description: Stable disease: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum LD since the treatment started.
  Progressive disease: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum of LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: Up to 112 days ( four 28-day cycles)
Population: All 18 participants were analyzed.
Measure: Number; unit: participants
Arm/Group | JI-101
Number analyzed (Participants) | 18
participants
  Cycle 2 - Stable Disease | 7
  Cycle 2 - Progressive Disease | 10
  Cycle 4 - Stable Disease | 5
  Cycle 4 - Progressive Disease | 2
  Cycle 6 - Stable Disease | 5
  Cycle 6 - Progressive Disease | 0
  Cycle 8 - Stable Disease | 3
  Cycle 8 - Progressive Disease | 2
  Cycle 10 - Stable Disease | 2
  Cycle 10 - Progressive Disease | 1
  Cycle 12 - Stable Disease | 2
  Cycle 12 - Progressive Disease | 0
  Cycle 14 - Stable Disease | 1
  Cycle 14 - Progressive Disease | 0
  Cycle 16 - Stable Disease | 1
  Cycle 16 - Progressive Disease | 0

4. Secondary Outcome: Days to Progression
Description: Progression: At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum of LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: Up to 112 days (four 28-day cycles) or longer if the patient is benefiting from treatment
Population: The efficacy analyses were performed using all patients, who had at least one post-treatment evaluation for tumor assessment (N=17). The overall response was based on the number of cycles of treatment before the participant experienced progressive disease.
Measure: Median (Full Range); unit: days
Arm/Group | All Subjects
Number analyzed (Participants) | 17
days | 55 [19 to 444]

ADVERSE EVENTS:
Time Frame: 2 years
Description: One subject was followed for an additional 5 months until the progression of disease.
Groups:
- JI-101: Maximum tolerated dose
Arm/Group | JI-101
Serious Adverse Events (participants affected / at risk) | 6/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JI-101 (N=18)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
peritonitis (Gastrointestinal disorders) | 1 (1)
metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
duodenal obstruction (Gastrointestinal disorders) | 1 (1)
impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
subarachnoid hemorrhage (Nervous system disorders) | 1 (1)
dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JI-101 (N=18)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Hyperacusis (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 4 (4)
Acquired corneal dystrophy (Eye disorders) | 1 (1)
Dellen (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 3 (3)
Eye pain (Eye disorders) | 1 (1)
Intraocular pressure increased (Eye disorders) | 2 (2)
Macular degeneration (Eye disorders) | 1 (1)
Pseudoexfoliation of lens capsule (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 3 (3)
Visual acuity reduced (Eye disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Abdominal tenderness (Gastrointestinal disorders) | 1 (1)
Aphthous stomatitis (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (9)
Oral pain (Gastrointestinal disorders) | 2 (2)
Pyrexia (Gastrointestinal disorders) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Tongue blistering (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7)
Asthenia (General disorders) | 2 (2)
Chills (General disorders) | 5 (5)
Edema peripheral (General disorders) | 1 (1)
Fatigue (General disorders) | 11 (11)
Feeling cold (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Mass (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 4 (4)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 4 (4)
Temperature intolerance (General disorders) | 1 (1)
Thirst (General disorders) | 1 (1)
Hyperbilirubinemia (Hepatobiliary disorders) | 2 (2)
Clostridial infection (Infections and infestations) | 2 (2)
Fungal infection (Infections and infestations) | 1 (1)
Furuncle (Infections and infestations) | 1 (1)
Nasal abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Vaginal abscess (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 2 (2)
Blood amylase decreased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood calcium decreased (Investigations) | 2 (2)
Blood chloride decreased (Investigations) | 1 (1)
Blood cortisol decreased (Investigations) | 1 (1)
Blood creatinine decreased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Blood glucose increased (Investigations) | 2 (2)
Blood potassium increased (Investigations) | 1 (1)
Blood pressure orthostatic (Investigations) | 1 (1)
Blood sodium decreased (Investigations) | 4 (4)
Blood uric acid increased (Investigations) | 1 (1)
Carbon dioxide decreased (Investigations) | 1 (1)
International normalized ratio increased (Investigations) | 3 (3)
Weight decreased (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 13 (13)
Dehydration (Metabolism and nutrition disorders) | 7 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 (1)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Dysgeusia (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 5 (5)
Hyperesthesia (Nervous system disorders) | 1 (1)
Hypoesthesia (Nervous system disorders) | 4 (4)
Migraine (Nervous system disorders) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Nightmare (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Incontinence (Renal and urinary disorders) | 1 (1)
Micturition disorder (Renal and urinary disorders) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Breast mass (Reproductive system and breast disorders) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sputum discolored (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3)
Heat rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5)
Night sweats (Skin and subcutaneous tissue disorders) | 5 (5)
Pain of skin (Skin and subcutaneous tissue disorders) | 4 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 (4)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin chapped (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Hot flush (Vascular disorders) | 9 (9)
Hypertension (Vascular disorders) | 10 (10)
Orthostatic hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No